CLINICAL TRIAL: NCT01693757
Title: Comparison of Functional Outcome Measures of Anterior Cruciate Ligament Reconstruction Using Either Patellar Tendon or Hamstring Tendon Grafts and Controls in Competitive Soccer Players: A Randomized Trial
Brief Title: Functional Outcome Anterior Cruciate Ligament Reconstruction
Status: Completed | Type: Observational
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Farshid Mohammadi, Director, University of Social Welfare and Rehabilitation Science
Other Study IDs: 3; USWR (Other: USWR)
Record Dates: First submitted 2012-05-25; First posted 2012-09-26 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Complications of Surgical Procedures or Medical Care
Keywords: Anterior Cruciate Ligament; Hamstrings versus patellar tendon; Hop test; Return to sports

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- BPTB group: Bone-patellar tendon-bone
- STG group: Semitendinosus and gracilis tendon
- Control: Healthy

SUMMARY:
The purpose of this study is to compare hop performance and jump landing strategy in soccer players with higher level sports activities after ACLR using either BPTB or STG and controls.

DETAILED DESCRIPTION:
The choice of graft for anterior cruciate ligament reconstruction (ACLR) remains controversial. Despite the need for outcome studies comparing bone-patellar tendon-bone (BPTB) with semitendinosus and gracilis tendon (STG), few studies have evaluated functional outcomes. The objective of the current study was to compare hop performance and jump landing strategy in soccer players with higher level sports activities after ACLR using either BPTB or STG and controls.

ELIGIBILITY:
Inclusion Criteria:

* ACLR and controls.

Exclusion Criteria:

* Musculoskeletal injuries

Ages: 21 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The patients with ACL deficiency were invited to participate in a randomized trial comparing ACLR with either a BPTB or STG graft.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2010-01; Primary Completion 2011-01 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Hop values for the both legs in Single, 6-m, Cross-over and Triple hops | Patients were followed up to 8 months post-surgery

SECONDARY OUTCOMES:
Landing and Take-off Ground Reaction Forces | Patients were followed up to 8 months post-surgery
Strength of Quadriceps and Hamstrings | Patients were followed up to 8 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mahyar Salavati, Professor, Study Director — USWR
Locations (1):
- USWR, Tehran, Iran